CLINICAL TRIAL: NCT00448240
Title: Erlotinib (Tarceva) Given Intermittently During First Line Standard Platinum Containing Chemotherapy for Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Erlotinib (Tarceva) During First Line Standard Platinum Containing Chemo for Advanced Squamous Cell Head and Neck Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low Accrual, Funding
Sponsor: Henry Ford Health System (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Haythem Ali, M.D., Senior Staff Physician, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HFHS 05-03
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Cancer; Carcinoma, Squamous Cell
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erlotinib (Experimental): Erlotinib (Tarceva) During First Line Standard Platinum Containing Chemo
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — loading dose of 300 mg on Day 2 followed by 150 mg daily Days 3 - 17 of each cycle of paclitaxel and cisplatin/carboplatin
  Other Names: Tarceva

SUMMARY:
The purpose of this study is to determine if combination Erlotinib, Cisplatin/Carboplatin, and Paclitaxel are effective first line treatment for metastatic, recurrent and persistent squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
We hypothesize that Erlotinib fails to enhance the effects of chemotherapy on response and survival because of Erlotinib's cytostatic effect, this results in a slowing down of the cell cycle, this in turn results in a hampering of the cytotoxic effect of chemotherapy leading to a lack of synergism with the combination. We propose that a sequential approach to the combination allows each drug to be used in its optimum time, by sequencing the Erlotinib, giving it 24 hours after chemotherapy we allow the chemotherapy to exert its effect with cells actively in cell cycle, but delivering the Erlotinib at a time when cells are trying to return to cell cycle hence slowing the growth rate of the tumor cell population. By withdrawing the Erlotinib about 4 days prior to the next chemotherapy cycle, we allow the cells to go back into cell cycle and therefore become susceptible to chemotherapy again.

Patients will be treated with intravenous paclitaxel over 3 hours followed by intravenous cisplatin/carboplatin on Day 1 of each 21 day cycle. Patients will be treated with Erlotinib at a loading dose of 300mg on Day 2 followed by 150 mg orally daily from Days 3-17 of each cycle of paclitaxel and cisplatin/carboplatin.

The primary objectives of this study are to assess the response rate of combination of erlotinib, cisplatin/carboplatin and paclitaxel in the first line treatment setting of metastatic, recurrent and persistent squamous cell carcinoma of the head and neck. Secondary objectives are to assess toxicity, median survival, and progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma of the head and neck region that is metastatic, recurrent or persistent after surgery and/or radiation
* No prior chemotherapy for metastatic, recurrent or persistent disease

Exclusion Criteria:

* Not more than 1 prior adjuvant or neoadjuvant chemotherapy regimen is allowed
* Chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haythem Ali, M.D/, Principal Investigator — Henry Ford Health System

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate of Intermittent Tarceva During First Line Standard Platinum Containing Chemotherapy
Description: Response rate of intermittent Tarceva will be measured by applying RECIST 1.0 criteria to measure response using radiologic testing.
Time Frame: Evaluated at 6-week intervals, up to an average of 18 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 6
Participants
  Disease Progression | 1
  Partial Response | 3
  Stable Disease | 2

ADVERSE EVENTS:
Arm/Group | Erlotinib
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=6)
lymphopenia (Blood and lymphatic system disorders) | 2
anemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
hearing loss (Ear and labyrinth disorders) | 1
lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenic fever (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
the study did not accrue fully and was closed due to poor accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No